CLINICAL TRIAL: NCT00756067
Title: A Study to Evaluate GSK Biologicals' Candidate Formulations of Pneumococcal Vaccines (GSK2189241A) in Elderly Subjects.
Brief Title: Evaluation of Pneumococcal Vaccine Formulations in Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111652
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Infections, Streptococcal
Keywords: Streptococcus pneumoniae; pneumococcal vaccine
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (7):
- Formulation 1 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189241A
- Formulation 2 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189241A
- Formulation 3 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189241A
- Formulation 4 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189241A
- Formulation 5 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189241A
- Formulation 6 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189241A
- 23 valent pneumococcal vaccine (Active Comparator)
  Interventions: Biological: Pneumo 23™

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK2189241A — Two doses of 0.5 ml will be administered intramuscularly; one dose at Month 0 and another at Month 2.
  Arms: Formulation 1; Formulation 2; Formulation 3; Formulation 4; Formulation 5; Formulation 6
Biological: Pneumo 23™ — One dose of 0.5 ml will be administered intramuscularly at Month 0, and a placebo dose to keep the blinding at Month 2.
  Arms: 23 valent pneumococcal vaccine

SUMMARY:
The purpose of this observer-blind study is to evaluate the safety, reactogenicity and immunogenicity of pneumococcal vaccines in elderly. Subjects will be vaccinated twice with an interval of two months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol should be enrolled in the study.
* Male or female subjects between, and including, 65 and 85 years old at the time of the first vaccination, in relatively stable health.
* Written informed consent obtained from the subject.

Exclusion Criteria:

* Previous vaccination against Streptococcus pneumoniae (with a licensed vaccine or with an investigational candidate vaccine).
* Vaccination with diphtheria/tetanus toxoids within one month preceding the first dose of study vaccine.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period or participation to another pharmaceutical/vaccine study.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of study vaccine, with the exception of the influenza vaccine which can be administered at least 7 days preceding or at least 7 days following any vaccine dose.
* Administration of immunoglobulins and/or any blood products within the last 3 months.
* Bacterial pneumonia within 3 years prior to 1st vaccination.
* Invasive pneumococcal disease (I.P.D) within 3 years prior to 1st vaccination.
* History of thrombocytopenia or bleeding disorder.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccine.
* History of administration of an experimental/licensed vaccine containing MPL or QS21.
* Current serious neurologic or mental disorders.
* Inflammatory processes such as known chronic active infections (e.g. Hepatitis B, C).
* All past or current malignancies (excluding non-melanic skin cancer) and lymphoproliferative disorders diagnosed or treated actively during the past 5 years.
* Acute disease at the time of enrolment.
* Physical examination positive for acrocyanosis, jaundice, splenomegaly
* Acute or chronic, clinically significant anaemia, pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by history, physical examination or laboratory screening tests at the discretion of the investigator.
* Laboratory evidence of haematological abnormalities.
* Laboratory evidence of biochemical abnormalities.
* History of chronic alcohol consumption and/or drug abuse.
* Other conditions that the principal investigator judges may interfere with study findings.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 168 (Actual)
Dates: Start 2008-09-19 (Actual); Primary Completion 2009-05-28 (Actual); Study Completion 2009-05-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of any vaccine related and grade 3 solicited local and general adverse events | During a 7-day follow up period after each vaccine dose
Occurrence of any vaccine related and grade 3 unsolicited adverse events | During a 31-day follow up period after each vaccine dose
Occurrence of any vaccine related serious adverse events (SAE) | From dose 1 to study conclusion
Occurrence of any grade 3 laboratory abnormalities | At 1 and 7 days after each vaccine dose

SECONDARY OUTCOMES:
Occurrence of any solicited local and general adverse events | During a 7-day follow up period after each vaccine dose
Occurrence of any unsolicited adverse events | During a 31-day follow up period after each vaccine dose
Occurrence of any laboratory abnormalities | At 1 and 7 days after each vaccine dose
Occurrence of any medically significant conditions prompting emergency room visits or physician visits regardless of casual relationship to vaccination or intensity | From dose 1 to study conclusion
Anti-pneumococcal and anti-NTHi candidate vaccine antigens | At Days 0, 30 and 90

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Sweden (3):
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Pauksens K, Nilsson AC, Caubet M, Pascal TG, Van Belle P, Poolman JT, Vandepapeliere PG, Verlant V, Vink PE. Randomized controlled study of the safety and immunogenicity of pneumococcal vaccine formulations containing PhtD and detoxified pneumolysin with alum or adjuvant system AS02V in elderly adults. Clin Vaccine Immunol. 2014 May;21(5):651-60. doi: 10.1128/CVI.00807-13. Epub 2014 Mar 5. PMID 24599529
- See also: Results for study 111652 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/111652?search=study&b%22b''%22#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register